CLINICAL TRIAL: NCT00052728
Title: A Phase II Trial Of Tipifarnib (R15777, ZARNESTRA) In Combination With Tamoxifen In Subjects With Metastatic Breast Cancer
Brief Title: Tipifarnib Plus Tamoxifen in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258720; NCI-03-C-0037; NCI-5540; NCT00048867 (obsolete NCT alias)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2005-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; tipifarnib

INTERVENTIONS:
Drug: tamoxifen citrate
Drug: tipifarnib

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Tamoxifen may fight breast cancer by blocking the use of estrogen. Combining tipifarnib with tamoxifen may be effective treatment for metastatic breast cancer.

PURPOSE: This phase II trial is studying how well giving tipifarnib together with tamoxifen works in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of tipifarnib administered with tamoxifen in women with hormone receptor-positive metastatic breast cancer (Phase I closed to accrual effective 10/23/2003).
* Determine the acute and chronic toxicity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the response rate and time to progression in patients treated with this regimen.

OUTLINE: This is an open-label study of tipifarnib (Phase I closed to accrual effective 10/23/2003). Patients are stratified according to benefit from prior hormonal therapy (yes vs no) (phase II).

* Phase I (closed to accrual effective 10/23/2003): Patients receive oral tipifarnib twice daily on days 1-21. Patients also receive oral tamoxifen daily on days 8-18 (during course I only) and on days 1-28 during all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Once the MTD is determined, additional patients are accrued and treated at that dose level in the phase II portion of the study.

Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 9-12 patients will be accrued for the phase I portion of this study (Phase I closed to accrual effective 10/23/2003). A total of 27-40 patients will be accrued for the phase II portion of this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic (stage IV) breast cancer
* Evidence of disease progression
* Measurable disease
* Must have been previously treated with at least 1 hormonal therapy with either an aromatase inhibitor or an estrogen receptor (ER)-modulating drug in the adjuvant or metastatic setting and meets 1 of the following criteria:

  * Hormone-responsive disease:

    * Stable disease (no recurrence or progression for at least 6 months)
    * Objective response
  * Hormone-nonresponsive disease:

    * No stable disease
    * No objective response
* Previously treated CNS disease allowed provided patient has a life expectancy of at least 3 months (phase I patients) (Phase I closed to accrual effective 10/23/2003)
* No CNS metastases (phase II patients)
* Hormone receptor status:

  * ER and/or progesterone receptor positive
* NOTE: As few as 1% positive cells considered positive

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* See Disease Characteristics

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL (unless evidence of Gilbert's disease)
* SGOT and SGPT less than 3 times upper limit of normal (unless liver involvement by tumor)

Renal

* Creatinine no greater than 1.5 mg/dL

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for 2 months after study participation
* No medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 2 prior chemotherapy regimens for metastatic disease (phase II patients)

  * No limitations on prior neoadjuvant or adjuvant regimens
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* See Disease Characteristics
* At least 6 months since prior tamoxifen
* Concurrent stable dose of steroids allowed (phase I patients) (Phase I closed to accrual effective 10/23/2003)

Radiotherapy

* No concurrent radiotherapy

Surgery

* Concurrent surgery allowed provided the need for surgery is not due to disease progression

Other

* Recovered from all prior therapy
* No prior warfarin
* No concurrent cytochrome p450-inducing anti-convulsants
* No other concurrent anticancer therapies
* Concurrent bisphosphonates for bone metastases allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnne Zujewski, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Result] Lebowitz PF, Eng-Wong J, Widemann BC, Balis FM, Jayaprakash N, Chow C, Clark G, Gantz SB, Venzon D, Zujewski J. A phase I trial and pharmacokinetic study of tipifarnib, a farnesyltransferase inhibitor, and tamoxifen in metastatic breast cancer. Clin Cancer Res. 2005 Feb 1;11(3):1247-52. PMID 15709195
- [Result] Lebowitz PF, Eng-Wong J, Balis F, et al.: A phase I trial of tipifarnib, a farnesyltransferase inhibitor, and tamoxifen in hormone-receptor positive metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 22 (Suppl 14): A-644, 38s, 2004.